CLINICAL TRIAL: NCT02382874
Title: Allogenic Adipose Derived Mesenchymal Stromal Cells Transplantation to Improve Kidney Function in Refractory Primary Nephrotic Syndrome (Focal Segmental Glomerulosclerosis,FSGS) ,a Phase I Clinical Trial
Brief Title: Allogenic AD-MSC Transplantation in Idiopathic Nephrotic Syndrome (Focal Segmental Glomerulosclerosis)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Kidney-005
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: Idiopathic nephrotic syndrome; adipose derived mesenchymal stromal cell; Focal segmental glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid | interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AD-MSC (Experimental): The patients with FSGS who underwent intravenous injection of AD-MSC.
  Interventions: Biological: Intravenous injection

INTERVENTIONS:
Biological: Intravenous injection — Intravenous injection of AD-MSC to the patients with FSGS

SUMMARY:
Idiopathic Focal Segmental Glumero Sclerosis (FSGS) is not very common but important manifestation of kidney disease.

FSGS has poor prognosis among the patterns of Idiopathic Nephrotic Syndrome (INS).

Even with treatment (Steroid therapy and cytotoxic immunosuppressant therapy), many patients eventually still require dialysis.

Cell therapy is useful in treatment of INS and mesenchymal stromal/stem cell is one of the cells that useful in the treatment of glomerulus disease.

Intravenous injection of allogeneic adipose derived mesenchymal stromal/stem cell will be done in 5 patients with refractory INS(FSGS). They will be followed 1, 2, 4 weeks and then monthly until a year following injection day.

DETAILED DESCRIPTION:
Primary FSGS thought to be a part of the immune-mediated disease. Main challenge is to decrease protein excretion in urine. Only 30% of children with FSGS achieve complete remission with steroids and other 30-40% patients experience remission (partial and complete) with cytotoxic immunosuppressant drugs. Even with these treatments, many patients eventually still require dialysis. Other treatment strategy doesn't exceed beyond symptomatic treatment and delaying the progression. Also risk of recurrence after kidney transplantation is 20-50%.

Cell therapy is one of the treatment strategies and mesenchymal stromal/stem cell is one modality that notice in glomerulus disease.

We will evaluate safety and efficacy of intravenous injection of allogeneic AD-MSC (adipose-derived mesenchymal stromal cell) in 5 refractory INS patients.They will be followed 1, 2, 4 weeks and then monthly until a year following injection day.

ELIGIBILITY:
Inclusion Criteria:

- Age 2-14 years at onset of signs or symptoms of FSGS 2- Primary FSGS involving either native kidneys or primary FSGS recurring after renal transplantation. Biopsy confirmed as primary FSGS (including all subtypes).

3-Estimated GFR ≥ 25 ml/min/1.73 m2 4- Up/c > 1.0 (g protein/g creatinine) on first am void 5- Steroid and IS resistance as defined by primary physician (patients with little or no reduction in protein excretion at 12 to 16 weeks are considered to be steroid resistant --A relapse is return of proteinuria to ≥3.5 g/day in someone who had undergone a complete or partial remission- IS resistance: no response to IS in 8-12 weeks) 6-At least one month from last immunization received has passed 7- Ability to understand and willingness to sign consent by patient legal guardian

Exclusion Criteria:

- 1- Are immunodeficient or have clinically significant chronic lymphopenia 2-Have an active infection or positive PPD test result 3-Have serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C infection 4-Have any complicating medical issues that interfere with study conduct or cause increased risk such as malignancies, systemic autoimmune disease, diabetes, blood disease, liver disease, etc.

5- Positive genetic mutation testing for WT1, Podocin, Nephrin

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Liver function | 2 weeks
  increase of liver enzymes 2 weeks after cell injection.
Serum creatinine | 2 weeks
  Decrease of serum creatinine 2 weeks after cell injection.
Proteinuria | 12 hour
  Reduction in proteinuria to <200 to 300 mg/day will be assessed by Changes in 24 hour urine protein analysis.

SECONDARY OUTCOMES:
Renal function | 12 hours
  will be assessed by change in serum levels of Cr, Urea and GFR. Time Frame: 12 hr after injection,1,2 weeks then monthly until a year after 1st injection.
Increase in anti inflammatory factors | 12 hours
  It will be assessed by change in serum levels of IL-2, 10. Time frame: 12 hour after injection then monthly until a year 1st injection.
Increase in Treg | 12hours
  It will be assessed by change in serum levels of Treg. Time frame: 12 hr after injection,1 week, 3, 6,12 months after 1st injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of department of regenerative medicine&cell therapy center,Royan Institute; Hassan Otukesh, MD, Study Director — Department Of Pediatric Nephrology and Dialysis, Ali aghar Children Hospital, Iran University of Medical Sciences, Tehran, Iran; Rozita Hosseini, MD, Principal Investigator — Department Of Pediatric Nephrology and Dialysis, Ali aghar Children Hospital, Iran University of Medical Sciences, Tehran, Iran; Soroosh Shekarchian, MD, Principal Investigator — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org